CLINICAL TRIAL: NCT04134494
Title: Effectiveness of Ablative Fractional 2940 nm Laser Treatment for Vulvar Lichen Sclerosus
Brief Title: Laser Treatment for Vulvar Lichen Sclerosus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was significantly impacted by the COVID-19 pandemic.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Sciton (Industry)
Responsible Party: Principal Investigator, Roger Lefevre, Instructor in Obstetrics, Gynecology and Reproductive Biology, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P000344
Record Dates: First submitted 2019-10-17; First posted 2019-10-22 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: Massachusetts residents
MeSH Terms: conditions — Vulvar Lichen Sclerosus | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: The objective was to enroll a single group of 30 patients with biopsy-proven Lichen sclerosus will be treated on a monthly basis for 3 months. Biopsy to be repeated at month #6. The biopsy from before treatment will be compared with biopsies after treatment. Enrollment ended early.
Masking Description: No masking will be used as all patients will receive the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): Women with biopsy-proven lichen sclerosus will be treated with the ProFractional hand piece using the sapphire plate stand-off (Sciton, Inc. Palo, Alto, CA). The laser energy is delivered in a scanning fractional pattern to ablate microchannels in tissue to allow faster healing. Treatment will be delivered in 3 sessions scheduled 4 weeks (+/- 1 week) apart
  Interventions: Device: Ablative Fractional 2940 nm Laser

INTERVENTIONS:
Device: Ablative Fractional 2940 nm Laser — * Treatment visit 1, month 0: On the first pass, the depth of the laser will be from 300 to 500 microns, or the thickness of 3 to 5 sheets of paper; the depth will be based on the biopsy that was used to diagnosis the lichen sclerosus. On the second pass, the depth will be 50 microns deeper than the first pass and the hand piece rotated 45˚.
  * Treatment visit 2, month 1: The first pass of the laser will be the same depth as the second pass from the last visit. The second pass will be 50 microns deeper and the hand piece rotated 45˚.
  * Treatment visit 3, month 2: The first pass of the laser will be the same depth as the second pass from the last visit. The second pass will be 50 microns deeper and the hand piece rotated 45˚.

SUMMARY:
The object of this non-randomized, prospective study is to assess the effectiveness of ablative fractional 2940 nm laser treatment of vulvar lichen sclerosus.

Aim 1: To assess physical and histological changes related to vulvar lichen sclerosus before and after laser treatment.

Aim 2: To evaluate participant satisfaction for laser treatment of vulvar lichen sclerosus.

The results of this study will determine whether fractional 2940 nm laser is an effective treatment option for lichen sclerosus, particularly for those participants not eligible for high-dose topical steroids or who have failed prior treatment with topical steroids.

DETAILED DESCRIPTION:
This will be a non-randomized, open-label, prospective study. Participants will be recruited in general and subspecialty obstetrics and gynecology clinics. Participants who meet all eligibility criteria, including providing written informed consent, will have three treatment visits and three follow-up visits in an outpatient setting. Participants will not be charged for any treatments.

At each treatment visit, participants will be asked to complete questionnaires to assess their symptoms. The investigators will also take photographs of the affected area at each treatment visit. Photographs will include only the area of lichen sclerosus, such that individuals cannot be identified in the photographs. Participant photographs will be taken using the BIDMC PhotoConsult iOS application that allows providers to upload photographs to a patient's online medical record through a secure application.

Women with biopsy-proven lichen sclerosus will be treated with the ProFractional hand piece using the sapphire plate stand-off (Sciton, Inc. Palo, Alto, CA). The laser energy is delivered in a scanning fractional pattern to ablate microchannels in tissue to allow faster healing. Treatment will be delivered in 3 sessions scheduled 4 weeks (+/- 1 week) apart.

Prior to receiving treatment, topical 4% lidocaine anesthetic will be applied to the affected area for 20-30 minutes and then wiped away. The treatment area will be cleaned and dried of any moisture prior to treatment. The disinfected standoff with sapphire plate will then be applied to the ProFractional hand piece. Based on the biopsy results, the appropriate ablation depth will be inputted with 11% treatment density selected. Each treatment will include two passes of the laser over the affected area.

* Treatment visit 1, month 0: On the first pass, the depth of the laser will be from 300 to 500 microns, or the thickness of 3 to 5 sheets of paper; the depth will be based on the biopsy that was used to diagnosis the lichen sclerosus. On the second pass, the depth will be 50 microns deeper than the first pass and the hand piece rotated 45˚.
* Treatment visit 2, month 1: The first pass of the laser will be the same depth as the second pass from the last visit. The second pass will be 50 microns deeper and the hand piece rotated 45˚.
* Treatment visit 3, month 2: The first pass of the laser will be the same depth as the second pass from the last visit. The second pass will be 50 microns deeper and the hand piece rotated 45˚.

Participants will return for follow-up visits at 1, 3, and 6 months (months 3, 6 and 9 of the study) following the third treatment.

* Follow-up visit 1, month 3

  * Participants will be asked to complete questionnaires to assess outcomes.
  * The investigators will take photographs of the affected area.
* Follow-up visit 2, month 6

  * Participants will be asked to complete questionnaires to assess outcomes.
  * The investigators will take photographs of the affected area.
  * Biopsy of area with lichen sclerosus; the biopsy will be done the same way as the one that was done to diagnosis your lichen sclerosus
* Follow-up visit 6, month 9

  * Participants will be asked to complete questionnaires to assess outcomes.
  * The investigators will take photographs of the affected area.

ELIGIBILITY:
We are currently recruiting Massachusetts residents only due to COVID-19.

Inclusion Criteria:

* Female
* Aged 18 years old or older
* Biopsy-proven active vulvar lichen sclerosus
* Characteristic changes of vulvar lichen sclerosus on gynecological exam
* Self-reported indication of one or more of the following symptoms of lichen sclerosus

  * Dryness
  * Itching
  * Burning
  * Bleeding
  * Blistering
  * Soreness
  * Easily bruises
  * Easily tears
  * Ulcerated lesions
  * Painful intercourse
* Ability to complete questionnaires in English
* Written, informed consent
* Willing and able to logistically follow schedule of treatments and follow-up visits

Exclusion Criteria:

* Receiving systemic immunosuppressant's (e.g. corticosteroids) within 4 weeks of enrollment
* Use of topical vulvar steroid-containing creams at the affected area within 4 weeks of enrollment
* Immunocompromised (e.g. lymphoma, AIDS, Wiskott-Aldrich syndrome)
* History of uncontrolled malignant disease
* Additional genital skin disease
* Known allergy or intolerance to topical anesthesia
* Known history of connective tissue disease
* Known propensity for keloid formations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Lefevre, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Women with biopsy-proven lichen sclerosus will be treated with the ProFractional hand piece using the sapphire plate stand-off (Sciton, Inc. Palo, Alto, CA). The laser energy is delivered in a scanning fractional pattern to ablate microchannels in tissue to allow faster healing. Treatment will be delivered in 3 sessions scheduled 4 weeks (+/- 1 week) apart
  Ablative Fractional 2940 nm Laser: • Treatment visit 1, month 0: On the first pass, the depth of the laser will be from 300 to 500 microns, or the thickness of 3 to 5 sheets of paper; the depth will be based on the biopsy that was used to diagnosis the lichen sclerosus. On the second pass, the depth will be 50 microns deeper than the first pass and the hand piece rotated 45˚.
  * Treatment visit 2, month 1: The first pass of the laser will be the same depth as the second pass from the last visit. The second pass will be 50 microns deeper and the hand piece rotated 45˚.
  * Treatment visit 3, month 2: The first pass of the laser will be the same depth as the second pass from the last visit. The second pass will be 50 microns deeper and the hand piece rotated 45˚.
Period: Overall Study
Arm/Group | Intervention
Started | 15
Completed | 13
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: 2 patients did not have the primary outcome assessed
Arm/Group | Intervention
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 patients did not have the primary outcome assessed
  Participants
    <=18 years | 0
    Between 18 and 65 years | 9
    >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants] — Self-reported sex collected on Study Questionnaire
  Participants
    Female | 13
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Baseline depth of lichen penetration [Median (Inter-Quartile Range); unit: Microns] — Baseline depth of penetration of Lichen sclerosus
  Microns | 600 [400 to 600]

OUTCOME MEASURES:

1. Primary Outcome: Change in Depth of Disease From Baseline to Three Months After the Last Laser Treatment
Description: The baseline depth of lichen sclerosus will be based on the results of the clinical biopsy performed before study participation. The investigators will use the study biopsy collected at the follow-up visit three months after the last treatment to determine resolution of disease or, if disease persists, to what depth. The biopsies will therefore serve as an objective means to determine effective treatment of disease.
Time Frame: From enrollment to 3 months after the last laser treatment
Population: Enrolled participants who had a post treatment biopsy
Measure: Median (Inter-Quartile Range); unit: microns
Groups:
- Intervention: The ProFractional hand piece using the sapphire plate stand-off (Sciton, Inc. Palo, Alto, CA) delivered laser energy in a scanning fractional pattern to ablate microchannels in tissue to allow faster healing. Treatment was be delivered in 3 sessions scheduled 4 weeks (+/- 1 week) apart
  Ablative Fractional 2940 nm Laser: • Treatment visit 1, month 0: On the first pass, the depth of the laser will be from 300 to 500 microns, or the thickness of 3 to 5 sheets of paper; the depth will be based on the biopsy that was used to diagnosis the lichen sclerosus. On the second pass, the depth will be 50 microns deeper than the first pass and the hand piece rotated 45˚.
  * Treatment visit 2, month 1: The first pass of the laser will be the same depth as the second pass from the last visit. The second pass will be 50 microns deeper and the hand piece rotated 45˚.
  * Treatment visit 3, month 2: The first pass of the laser will be the same depth as the second pass from the last visit. The second pass will be 50 microns deeper and the hand piece rotated 45˚.
Arm/Group | Intervention
Number analyzed (Participants) | 13
microns | 0 [-100 to 300]

2. Secondary Outcome: Change in Symptoms and Quality of Life Using the Vulvovaginal Symptom Questionnaire (VSQ)
Description: The VSQ is a 21-item written questionnaire with four scales: symptoms, emotions, life-impact, and sexual impact. Each item is assessed with yes or no questions. If a participant answers no, they receive a score of 0, and if the participant answers yes, they receive a score of 1 for each question. The results are added to a composite score.
  Minimum score (better outcome): 0 Maximum score (worse outcome): 21
Time Frame: From enrollment to 3 months after last laser treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | -3 [-4 to 0]

3. Secondary Outcome: Change in Symptoms Using the Patient Global Impression Scale of Change (PGIC)
Description: The PGIC is a written questionnaire to assess change in status or symptoms over time. Patients can say that their symptoms are: very much improved (1), much improved (2), minimally improved (3), no change (4), minimally worse (5), much worse (6) or very much worse (7).
  Minimum score (better outcome): 1 Maximum score (worse outcome): 7
Time Frame: 3 months after last laser treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 3 [2 to 3]

4. Secondary Outcome: Change in Symptom Severity Using the Patient Global Impression Scale of Severity (PGIS)
Description: The PGIs is a written questionnaire to assess current status or symptoms. Patients can say that their symptoms are: normal (1), mild (2), moderate (3), or severe (4).
  Minimum score (better outcome): 1 Maximum score (worse outcome): 4
Time Frame: From enrollment to 3 months after last laser treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 0 [-1 to 0]

5. Secondary Outcome: Satisfaction With Treatment Using a Participant Satisfaction Questionnaire
Description: Using a written questionnaire, patients will be asked how satisfied they were with the treatment. They can choose that they are extremely satisfied (1), somewhat satisfied (2), neither satisfied nor dissatisfied (3), somewhat dissatisfied (4), or extremely dissatisfied (5).
  Minimum score (better outcome): 1 Maximum score (worse outcome): 5
Time Frame: 3 months after last laser treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale | 2 [2 to 3]

ADVERSE EVENTS:
Time Frame: Baseline to six months
Description: Light spotting (bleeding from the area outside the vagina where the laser is used) Allergic reaction to topical anesthetic (numbing cream) Infection from the biopsy or the laser treatment
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=13)
Light spotting (Reproductive system and breast disorders) | 0 (0) — Bleeding from the area outside the vagina where the laser is used
Allergic reaction to topical anesthetic (Skin and subcutaneous tissue disorders) | 0 (0)
Infection from the biopsy or the laser treatment (Infections and infestations) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/94/NCT04134494/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04134494/ICF_002.pdf